CLINICAL TRIAL: NCT03700489
Title: Mycological Comparative Study Between Single Maxillary Denture Fabricated From Rapid Heat Cure Acrylic Resin Material and Conventional Acrylic Resin Material Modified by Titanium Dioxide Nanoparticles
Brief Title: Mycological Comparative Study on Maxillary Dentures of Two Different Materials
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ali ibrahim mahmoud shamardal (Other)
Responsible Party: Sponsor-Investigator, Ali ibrahim mahmoud shamardal, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Acrylic vs Tio2 reinforced
Record Dates: First submitted 2018-09-26; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Effect of Tio2 Nanoparticles on Candida Aggregation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients take titanium dioxide denture (Experimental): patients will receive titanium dioxide denture (made from conventional acrylic resin modified by titanium dioxide nanoparticles ) for 1 month in the initial phase of the trial then in the later phase after one month they will receive( rapid heat cured acrylic resin)denture
  Interventions: Other: titanium dioxide denture
- patients take rapid heat denture (Placebo Comparator): patients will receive rapid heat denture for 1 month in the initial phase of the trial then in the later phase patients will receive titanium dioxide denture (made from conventional acrylic resin modified by titanium dioxide nanoparticles )
  Interventions: Other: titanium dioxide denture

INTERVENTIONS:
Other: titanium dioxide denture — patients will receive titanium dioxide denture (made from acrylic resin with titanium dioxide nanoparticles ) for 1 month in the initial phase then in the second phase after one month they will receive( rapid heat cured acrylic resin)denture according to the principle of crossover des

SUMMARY:
Cross over design the investigator divide participants to two groups group (A) will receive rapid heat cured denture base material and group (b) will receive the acrylic denture modified by titanium dioxide nanoparticles and after washout period alternatively group (a) will receive the acrylic denture modified by titanium dioxide nanoparticles AND group (b) will receive rapid heat cured denture base material the investigator will take swaps from dentures to count the candida species

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous maxillary arch and partially dentate mandibular arch with adequate interarch space.
* The edentulous ridges should be covered by firm healthy mucosa.
* Angle class I maxillomandibular relation.
* Healthy and cooperative patient

Exclusion Criteria:

* Patients with bad habits as severe clenching or bruxism, drug or alcohol addiction, moderate or heavy smoking (greater than 10 cigarettes per day).
* Previous history of radiotherapy or chemotherapy.
* Any skeletal problem dictates surgical intervention

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2018-10-20 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Mycological investigation | 6 months
  Count of candida on the fitting surface of denture by (CFU) unit

IPD SHARING:
Plan to Share IPD: Undecided